CLINICAL TRIAL: NCT01320306
Title: Intracranial Aneurysms and Cognitive Function
Status: Terminated | Type: Observational
Why Stopped: Could not be implemented
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/2292-2
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2012-05

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Subarachnoid hemorrhage: A group of patients suffering aneurismal subarachnoid hemorrhage will participate in a fMRI study.
- Prophylactic surgical treatment of un-ruptured aneurysms: A retrospective follow-up study of patients who have received prophylactic surgical treatment of un-ruptured aneurysms
- Conservative treatment: A retrospective follow-up of patients receiving conservative (life stile etc.) treatment of un-ruptured aneurysms.
- Control group of healthy subjects: Control group of healthy subjects

SUMMARY:
The prevalence rate of intracranial aneurysms in the adult population is close to 5%. Rupture risk of such aneurysms causing subarachnoid hemorrhage (SAH) can be substantial.Most patients suffering from an aneurysmal SAH are in their mid life, i.e., 30 to 60 years old. Aneurysmal SAH may cause disability and mortality. The present study includes a follow-up study and a cross-sectional fMRI study. The purpose of the follow-up study is to monitor patients receiving prophylactic surgical treatment of their un-ruptured aneurysms to examine whether such treatment is associated with cognitive, psychosocial and/or neurologic sequela. The purpose of the cross-sectional fMRI study is to examine the relationship between memory function and brain activity among SAH patients. Memory impairment is often found among aneurysmal SAH patients. Using fMRI can possibly shed some light on whether such memory impairment may be caused by diffuse cerebral damage or a focal damage at the aneurysm site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with un-ruptured aneurysms in the anterior communicating artery and the middle cerebral artery.
* A subgroup of patients suffering aneurismal subarachnoid hemorrhage.

Exclusion Criteria:

* History of earlier cerebrovascular, psychiatric or neurological disease.
* Age older than 75 years
* Lack of fluency in Norwegian
* Alcohol or Substance abuse
* Aphasia
* Substantial vision or hearing deficits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with un-ruptured aneurysms in the anterior communicating artery and the middle cerebral artery.A subgroup of patients suffering aneurismal subarachnoid hemorrhage.
  University Hospital of North Norway
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-01-31 (Actual); Study Completion 2012-01-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Each subject will undergo one assessment of cognitive function. The assessment lasts about 2.5 hours including breaks.
  Neuropsychological Assessment

SECONDARY OUTCOMES:
Neurological status | Each subject will undergo one clinical assessment of neurological status.
  A clinical examination of neurological status
fMRI | A subgroup of patients will participate in a fMRI study once
  A subgroup of patients will participate in a fMRI study once

CONTACTS AND LOCATIONS:
Overall Officials: Tor Ingebrigtsen, Phd, Study Chair — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Background] Isaksen JG, Bazilevs Y, Kvamsdal T, Zhang Y, Kaspersen JH, Waterloo K, Romner B, Ingebrigtsen T. Determination of wall tension in cerebral artery aneurysms by numerical simulation. Stroke. 2008 Dec;39(12):3172-8. doi: 10.1161/STROKEAHA.107.503698. Epub 2008 Sep 25. PMID 18818402
- [Background] Sandell T, Isaksen J, Bajic R, Ingebrigtsen T. [Treatment of intracranial aneurysms]. Tidsskr Nor Laegeforen. 2005 Aug 25;125(16):2188-91. Norwegian. PMID 16138132